CLINICAL TRIAL: NCT05914558
Title: Comorbid Painful Temporomandibular Disorder Among Trigeminal Neuralgia Patients
Brief Title: Comorbid Painful TMD Among Trigeminal Neuralgia
Acronym: TNTMD
Status: Withdrawn | Type: Observational
Why Stopped: Due to lack of funding, we have been unable to continue research activities. The future related to funding support does not look promising, therefore it is best to discontinue this project.
Sponsor: University of Minnesota (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: UMN IRB No. 00008873; JHU IRB No. 00388974 (Other: John Hopkins Univeristy)
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Trigeminal Neuralgia; Temporomandibular Disorder; Myofascial Pain; Trigeminal Neuropathy
MeSH Terms: conditions — Trigeminal Neuralgia; Temporomandibular Joint Disorders; Trigeminal Nerve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TN cohort: The patient was diagnosed with trigeminal neuralgia which has active symptoms in the past 30 days.
  Interventions: Diagnostic Test: Clinical appointment

INTERVENTIONS:
Diagnostic Test: Clinical appointment — One clinical interview and examination to confirm the diagnosis of trigeminal neuralgia and temporomandibular disorder.

SUMMARY:
An observational study following up with trigeminal neuralgia patients to understand their comorbid facial pain condition, specifically temporomandibular disorder.

DETAILED DESCRIPTION:
This multi-center prospective observational cohort study aims to investigate the prevalence of comorbid Temporomandibular disorders (TMD) among trigeminal neuralgia (TN) patients. Trigeminal neuralgia patients with active TN status from three clinical sites (University of Minnesota, School of Dentistry, Orofacial Pain Clinic; Mhealth Fairview, Clinical Surgical Center, Neurosurgery Clinic; John Hopkins University, Anesthesiology, and Critical Care Clinic) could enroll in this study voluntary. All the patients will be evaluated by a provider using standard clinical assessment for TN and TMD, along with validated RedCap questionnaires for TN and TMD diagnosis, and be followed up every six months for 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients visited the three clinical sites for facial pain
* Patients diagnosed with trigeminal neuralgia
* Has active pain symptoms in the past 30 days

Exclusion Criteria:

* Non-English speakers
* Patients with psychiatric disorders that might alter pain perception
* Adults lack the capacity to provide informed consent.
* Persons under the age of 18.
* All vulnerable populations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that visited three clinical centers in the study who sought care for their facial pain were diagnosed with trigeminal neuralgia, with active symptoms in the past 30 days.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence | 2 years
  Prevalence of comorbid painful TMD among TN patient

SECONDARY OUTCOMES:
Diagnostic questionnaire | 2 years
  The sensitivity, specificity of the diagnostic questionnaire for TN and TMD

CONTACTS AND LOCATIONS:
Overall Officials: Donald Nixdorf, DDS,MS, Principal Investigator — University of Minnesota; Qiman Gao, DDS,MS,PhD, Study Director — University of Minnesota
Locations (2):
- United States (2):
  - John Hopkins University, Baltimore, Maryland
  - University of Minnesota, Department of Neurosurgery, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
The final results will be shared with all the participants as a summary.
Supporting Information: CSR
Time Frame: By end of 2024